CLINICAL TRIAL: NCT00823199
Title: An Open Trial of Allopurinol in Patients With Poorly Responsive Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bronx Psychiatric Center (Other Government)
Responsible Party: Principal Investigator, Nigel Bark MD, Director Schizophrenia Research, Bronx Psychiatric Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICFV12/02
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allopurinal treatment (Experimental): Allopurinal 300mg once daily by mouth for four weeks
  Interventions: Drug: Allopurinal

INTERVENTIONS:
Drug: Allopurinal — 300mg once daily by mouth for four weeks

SUMMARY:
This is a four week open label trial of ALLOPURINOL to the treatment regime of ten (10) poorly responsive patients with schizophrenia, monitoring their response and side-effects. No change in medication is required.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with schizophrenia and poor response (no prospect of discharge because of symptoms)

Exclusion Criteria:

* Over 65
* Renal or liver disease
* Diabetes
* Hypertension
* Taking thiazides or ACE inhibitors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Bark, MD, Principal Investigator — Bronx Psychiatric Center

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten subjects were recruited, in-patients in a State Hospital, between 2005 and 2008
Period: Overall Study
Arm/Group | Allopurinal Treatment
Started | 10
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Group 1: All participants
Arm/Group | Group 1
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) Measures Symptoms of Schizophrenia
Description: Symptom scale Score 30 (best, no symptoms of schizophrenia) to 210 (worst)
Time Frame: baseline and 4 weeks
Population: Two subjects withdrew before the first week's evaluation
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Allopurinal Treatment
Number analyzed (Participants) | 8
scores on a scale
  Baseline | 95 (22)
  End | 75 (17)

2. Secondary Outcome: Simpson Angus Scale for Parkinsonism
Description: Measures drug induced parkinsonism, score 0 (best, no Parkinsonism) to 36 (worst)
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Allopurinal Treatment
Number analyzed (Participants) | 8
score on scale
  Baseline | 0.37 (0.74)
  End | 1.75 (3.1)

3. Post Hoc Outcome: Uric Acid Level
Time Frame: Baseline and 4 weeks
Population: 2 subjects had missing data
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Allopurinal Treatment: all participants
Arm/Group | Allopurinal Treatment
Number analyzed (Participants) | 6
mg/dL
  Baseline | 5.9 (1.7)
  End | 3.8 (0.7)

ADVERSE EVENTS:
Time Frame: During the 4 week study
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No